CLINICAL TRIAL: NCT03611543
Title: Evaluating Image Quality and Comfort of an Investigational Curved Paddle Compared to a Standard Paddle
Status: Completed | Type: Observational
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-03
Record Dates: First submitted 2016-10-20; First posted 2018-08-02 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Tomosynthesis; 3D Mammogram; Diagnostic Mammogram
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- STANDARD OF CARE: All the subjects enrolled in this study will be under a routine screening mammogram or undergoing a diagnostic mammogram using the standard of care (SOC) flat paddle.
  The Universal Pain Assessment Tool (UPAT) will be used to determine the comfort perception of each subject with the SOC paddle. The UPAT ranges from 0 to 10, where 0 represents 'no pain' and 10 'worst pain possible'.
  Interventions: Device: Standard of Care Flat Paddle
- INVESTIGATIONAL: All the subjects enrolled in this study will be under a routine screening mammogram or undergoing a diagnostic mammogram using the investigational (INV) curved paddle.
  The Universal Pain Assessment Tool (UPAT) will be used to determine the comfort perception of each subject with the INV paddle. The UPAT ranges from 0 to 10, where 0 represents 'no pain' and 10 'worst pain possible'.
  Interventions: Device: Investigational Curved Paddle

INTERVENTIONS:
Device: Standard of Care Flat Paddle — X-Ray Mammogram Exam.
  Each screening subject will receive a 4-view 2D plus 3D combination imaging: Left Cranial Caudal (LCC), Left Medial Oblique (LMO), Right Cranial Caudal (RCC), and Right Medial Oblique (RMLO) with the current standard of care (SOC) flat paddle.
  Each diagnostic subject will have her prescribed diagnostic 2D plus 3D combination imaging (CC or MLO) with the SOC flat paddle. The image view (CC or MLO) will be based on the visibility of the area of interest for which the diagnostic imaging was ordered.
  The amount of compression applied in all mammograms will be to achieve tautness.
  Groups: STANDARD OF CARE
Device: Investigational Curved Paddle — X-Ray Mammogram Exam.
  Each screening subject will receive a CC and an MLO in one of her breasts as determined by a randomization scheme with the investigational (INV) curved paddle.
  Each diagnostic subject will have her prescribed diagnostic 2D plus 3D combination imaging (CC or MLO) with the INV curved paddle. The image view (CC or MLO) will be based on the visibility of the area of interest for which the diagnostic imaging was ordered.
  The amount of compression applied in all mammograms will be to achieve tautness.
  Groups: INVESTIGATIONAL

SUMMARY:
The goal of this study is to evaluate patient comfort during compression with a standard flat mammographic paddle and an investigational curved paddle. This is a study that will be performed with x-ray imaging and will be used to determine if an overall reduction in pain can be appreciated in patients without loss in image quality as compared to the current standard mammogram. Another benefit of the curved paddle may be an increase of perceivable and measurable tissue capture.

DETAILED DESCRIPTION:
The study will be conducted in the United States at up to 5 centers. The study will enroll up to 600 subjects. The number of subjects was chosen to allow evaluation of screening and diagnostic patients with a variety of breast densities (fatty, scattered densities, heterogeneously dense or extremely dense) and women with a range of breasts sizes that fit on the current detector. The evaluation of pain reduction will be the primary endpoint, while examining the potential of increased tissue capture without a compromise in image quality will be assessed as secondary endpoints. The enrollment will be consecutive for subjects who sign informed consent to participate. Women participating in the study will present for a screening or diagnostic imaging exam.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female of any race and ethnicity
* Screening Subject is at least 40 years old, Diagnostic subjects are at least 25 years old
* Subject will be referred for a screening or a diagnostic work-up with tomosynthesis as part of the exam

Exclusion Criteria:

* Subjects who are pregnant or who think they may be pregnant
* Subjects lactating or presenting with discharge
* Women too large for the detector
* Subjects who cannot give informed consent

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women participating in the study will present for a screening or diagnostic imaging breast exam.
Sampling Method: Non-Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Waqas, Study Director — Hologic, Inc.
Locations (4):
- United States (4):
  - Stamford Hospital, Stamford, Connecticut
  - Elizabeth Wende Breast Clinic, Rochester, New York
  - Solis Mammagroaphy, Addison, Texas
  - TOPS Comprehensive Breast Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited based on inclusion/exclusion criteria from protocol 16-03 at 4 clinical sites between October 2016 and June 2018.
Pre-assignment Details: This study involved subjects undergoing a mammogram exam (screening or diagnostic).
  All subjects were X-ray imaged using the standard of care (SOC) flat paddle and the investigational (INV) curved paddle. Thus, the subjects in the SOC group were the same as those in the INV group.
  A total of 443 subjects were initially enrolled. Of those, 14 did not complete the study.
Units Other Than Participants: Mammogram exams in total
Groups:
- Standard of Care Flat Paddle: Subjects involved in this study underwent a screening routine mammogram or a diagnostic mammogram using the standard of care (SOC) flat paddle.
  A screening mammogram involved 4-image views (both breasts: LCC, LMO, RCC, RMLO) with the SOC paddle.
  A diagnostic mammogram involved 2-image views (CC and MLO) of the breast of interest with the SOC paddle.
- Investigational Curved Paddle: Subjects involved in this study underwent a screening routine mammogram or a diagnostic mammogram using the investigational (INV) curved paddle.
  A screening mammogram involved 2-image views (CC and MLO) in one of the breasts as determined by a randomization scheme.
  A diagnostic mammogram involved 2-image views (CC and MLO) of the breast of interest only.
Period: Overall Study
Arm/Group | Standard of Care Flat Paddle | Investigational Curved Paddle
Started | 443; 443 Mammogram exams in total | 443; 443 Mammogram exams in total
Completed | 429; 429 Mammogram exams in total | 429; 429 Mammogram exams in total
Not Completed | 14; 14 Mammogram exams in total | 14; 14 Mammogram exams in total
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Device failure | 2 | 2
Not completed — Missing information | 5 | 5

BASELINE CHARACTERISTICS:
Population: This study involves subjects undergoing a mammogram exam (screening or diagnostic).
  These subjects were X-ray imaged using the SOC and INV paddles to determine changes in their comfort level and establish a direct comparison between devices.
  This means the subjects in the SOC group are the same as those in the INV group.
  This section consolidates (combines) all the subjects enrolled as one group rather than two groups because we're evaluating both devices on the same subjects.
Groups:
- All Enrolled Subjects: This study involves subjects undergoing a mammogram exam (screening or diagnostic).
  These subjects were X-ray imaged using the SOC and INV paddles to determine changes in their comfort level and establish a direct comparison between devices.
  This means the subjects in the SOC group are the same as those in the INV group.
  This section consolidates (combines) all the subjects enrolled as one group rather than two groups because we're evaluating both devices on the same subjects.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 429
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Subjects analyzed based on complete data set availability
  years | 54.6 (11)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Subjects analyzed based on complete data set availability
  Participants
    Female | 429
    Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 374
  African American/Black | 29
  Hispanic/Latino | 20
  Asian | 2
  Indian/Persian | 3
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 429
BI-RADS Breast Density Assessment [Number; unit: participants]
  Type A (Breasts are almost entirely fatty) | 47
  Type B (Breasts are mainly fatty, with some scattered areas of dense tissue) | 192
  Type C (Breasts are a mixture of fatty and dense tissue) | 147
  Type D (Breasts are almost entirely dense) | 31
  Blank (No breast density category was recorded for the subjects) | 12

OUTCOME MEASURES:

1. Primary Outcome: Subject Comfort
Description: The Universal Pain Assessment Tool (UPAT) was used to assess each subject's comfort perception with each paddle (SOC and INV).
  The UPAT ranges from 0 to 10, where 0 represents 'no pain' and 10 'worst pain possible'.
Time Frame: 1 day (Day of procedure, No follow-up)
Population: The number of participants analyzed per group differs from the number provided in the Participant Flow module (429).
  Two subjects' pain scores were unclear when imaged with the INV paddle. For this reason, the analysis was done by contemplating 427 subjects.
  Three subjects' pain scores were unclear when imaged with the INV paddle. For this reason, the analysis was done by contemplating 426 subjects.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- INVESTIGATIONAL: All the subjects enrolled in this study will be under a routine screening mammogram or undergoing a diagnostic mammogram using the investigational (INV) curved paddle.
- STANDARD OF CARE: All the subjects enrolled in this study will be under a routine screening mammogram or undergoing a diagnostic mammogram using the standard of care (SOC) flat paddle.
Arm/Group | INVESTIGATIONAL | STANDARD OF CARE
Number analyzed (Participants) | 427 | 426
score on a scale | 2.6 [2.3 to 2.6] | 4.0 [3.6 to 4.1]
Statistical Analysis 1: Comparison: INVESTIGATIONAL vs STANDARD OF CARE; Test type: Superiority; p < 0.0001, Wilcoxon Rank-Sum test — Information related to the INVESTIGATIONAL group

2. Secondary Outcome: Breast Tissue Coverage
Description: An expert technologist evaluated the performance of the SOC and the INV paddles in 388 subjects.
  For each participant, the technologist answered which paddle was better at pulling in more breast tissue during imaging between SOC and INV (all subjects were imaged with both paddles during the same session).
  The technologist rated the paddles using a 5-point Likert scale, where -2 and -1 values mean that the SOC paddle performed better or slightly better, 0 means equal performance between paddles, and 2 and 1 mean that the INV performed better or slightly better than the SOC paddle.
  Note that different technologists were involved in the image acquisition. An acceptable tissue coverage for this study refers to having sufficient breast tissue (a balance between fatty and glandular tissue) in the image acquired so that any potential abnormalities can be effectively identified.
Time Frame: 1 Day (Day of procedure, No Follow-up)
Population: The number of participants analyzed per group differs from the number provided in the Participant Flow module (429).
  Technologists did not provide an answer to the question about preference for tissue coverage in 41 cases. For this reason, the analysis was done in 388 subjects only.
  The same 388 subjects are part of both groups: INV and SOC groups. Therefore, the results are shown combined in the data table.
Measure: Count of Participants; unit: Participants
Groups:
- All Enrolled Subjects: Participant subjects were imaged (X-ray imaging of breast tissue) using the investigational (INV) curved paddle and the standard of care (SOC) flat paddle. After this process, the technologist in charge of image acquisition reported performance preference between paddles in terms of tissue coverage. If equal breast tissue was pull in with both paddles, this was also reported.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 388
Participants
  Rate -2 or -1 (SOC better or slightly better than INV) | 69
  Rate 0 ( SOC equal INV) | 162
  Rate 2 or 1 ( INV better or slightly better than SOC) | 157

3. Secondary Outcome: Overall Determination of Image Quality
Description: An expert radiologist reviewed, side by side, 3D images acquired with the INV and the SOC paddles in 420 subjects.
  The radiologist rated the images using a 5-point Likert scale, where -2 and -1 values mean that the images acquired with the SOC paddle have better or slightly better quality, 0 means equal quality between the images, and 2 and 1 mean that the images acquired with the INV paddle have better or slightly better quality than the SOC paddle.
  To determine overall clinical image quality or image acceptability, the radiologist considered whether the images reviewed have fair lesion visibility (when a lesion is present), good breast tissue separations of structures, good breast tissue coverage, no artifacts due to patient motion, and can be used to determine breast tissue density.
  Note that not all the 420 images were reviewed by the same radiologist.
Time Frame: 1 day (Day of procedure, No Follow-up)
Population: The number of participants analyzed per group differs from the number provided in the Participant Flow module (429).
  Data results related to image quality were unclear in nine subjects. For this reason, the analysis considered only 420 subjects.
  These 420 subjects are the same in both groups, INV and SOC, so the images can be comparable.
  Therefore, the results shown are combined in the data table.
Measure: Count of Participants; unit: Participants
Groups:
- All Enrolled Subjects: Screening and Diagnostic subjects were imaged (X-ray imaging of breast tissue) using the INV curved paddle and the SOC flat paddle. After this process, an expert radiologist compared the images, side by side, and reported preference in terms of overall image quality between INV and SOC. Equal image quality between images was also reported.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 420
Participants
  Rate -2 or -1 (SOC better or slightly better than INV) | 27
  Rate 0 (SOC equal INV) | 330
  Rate 2 or 1 (INV better or slightly better than SOC) | 63

ADVERSE EVENTS:
Time Frame: 1 day (Day of procedure, No follow-up)
Description: For this study, the subjects in the SOC group are the same as those in the INV group.
  All subjects were combined in a single group for the adverse event reporting because we're evaluating both devices on the same subjects.
Groups:
- All Enrolled Subjects: This study involves subjects undergoing a screening mammogram or diagnostic exams.
  These subjects were imaged using the SOC and INV paddles to determine changes in their perception of comfort and establish a valid comparison.
  The subjects in the SOC group are the same as those in the INV group. For this reason, the subjects were consolidated as one group, which involved all the subjects enrolled in the study.
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/429
Serious Adverse Events (participants affected / at risk) | 0/429
Other Adverse Events (participants affected / at risk) | 0/429

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03611543/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03611543/ICF_001.pdf